CLINICAL TRIAL: NCT02222519
Title: Interaction of Statins and Nondepolarizing Muscle Relaxants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huang-wei LV (Other)
Responsible Party: Sponsor-Investigator, Huang-wei LV, Professor, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Other Study IDs: 2014071801
Record Dates: First submitted 2014-08-14; First posted 2014-08-21 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Pain
Keywords: statins; nondepolarizing muscle relaxants; rocuronium; myalgia
MeSH Terms: conditions — Pain; Myalgia | interventions — Rocuronium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Statin use group: patients taking statins for at least 3 months
  Interventions: Drug: Rocuronium
- non statin use: no history of taking statin
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — Rocuronium 0.6mg/kg iv single dose
  Other Names: Rocuronium Bromide Injection; Esmeron; http://www.msdchina.com.cn/

SUMMARY:
provide evidence for prevention or reduction muscle pain.

DETAILED DESCRIPTION:
The purpose of this study is to determine interaction of statins and nondepolarizing muscle relaxant,In order to provide evidence for prevention or reduction muscle pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists physical status I-III
* Patients taking statins for at least 3 months and those who had never used statins were considered to be eligible

Exclusion Criteria:

* Orthopedic
* Spinal surgery
* Surgery involving extensive muscle manipulation
* History of liver and kidney failure
* Neuromuscular disease
* Susceptibility to or family history of malignant hyperthermia
* Extensive denervation of skeletal muscle
* Chronic pain syndromes
* Taking medications that might interact with the effect of rocuronium or serum myoglobin difficult intubation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients taking simvastatin, lovastatin, atorvastatin, or pravastatin for at least three months.
  Patients not taking simvastatin, lovastatin, atorvastatin, or pravastatin for at least three months
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
plasma myoglobin concentration | 20 minutes after administration

SECONDARY OUTCOMES:
muscle pain | 2 and 24 hours postoperatively
serum potassium concentration | 2 and 24 hours postoperatively
plasma creatine phosphokinase concentration | 2 and 24 hours postoperatively
urine myoglobin and onset plus duration of succinylcholine block | 2 and 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Huangwei Lv, Professor, Study Director — the Anesthesiology Department
Locations (1):
- China Medical University, Shenyang, Liaoning, China